CLINICAL TRIAL: NCT00247832
Title: Readiness for Discharge Following Lobectomy: Effects of the Thoracic Risk Intervention and Management (T.R.I.M.) Protocol
Brief Title: Readiness for Discharge Following Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C05 - 0500
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Pain; Anxiety
Keywords: Monitoring, early mobilization, motivation modality, visitation rate, step rates, anxiety, pain; Elective lobectomy
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention)
- 2 (Experimental): Self-directed motivation
  Interventions: Behavioral: Self-directed motivation
- 3 (Experimental): Personal motivational interviewing
  Interventions: Behavioral: Personal motivational interviewing

INTERVENTIONS:
Behavioral: Self-directed motivation — Post-lobectomy patients are provided with a booklet that outlines expected physical activities (sitting up, walking arm exercises) to aim for each day after surgery. It also provides room for the patients to record what they have accomplished.
  Arms: 2
Behavioral: Personal motivational interviewing — Post-lobectomy patients receive daily visits from a study coordinator aimed to motivate the patient to complete various physical activities each day after surgery. The study coordinator goes through the same booklet that is given to Group 2 and helps patients set goals and record their accomplishments.
  Arms: 3

SUMMARY:
This study aims to examine the relationship between the patient's perception of readiness for discharge after lobectomy and mobilization rates, frequency of visitation by family and friends, anxiety levels and pain levels. We will test the hypotheses that a) those patients who walk farther early after surgery and who have more visitors and decreased anxiety and pain levels will have a greater self-perceived readiness for discharge and b) that patients who receive daily ambulation goals and personal motivation will have higher step rates, and therefore have a greater self-perceived readiness for discharge, than those that do not. We will monitor patients, during the post-operative recovery period using pedometers to count steps taken, visitor log sheets, and questionnaires on the patients' anxiety, pain and perceived readiness for discharge. Furthermore, we will examine how the patient's self-perceived readiness for discharge is affected by study interventions which include ambulation goals and daily personal motivation.

DETAILED DESCRIPTION:
There is currently little information on indicators and factors of a patient's readiness for discharge. Vancouver General Hospital is attempting to create a standardized clinical pathway for individuals who have undergone a lobectomy, to increase patient satisfaction and decrease hospital stay and complication rates. This study aims examine the relationship between the patient's readiness for discharge after lobectomy and their mobilization rate (measured as the number of steps taken in a day), frequency of visitation by family and friends, the level of anxiety and the level of pain experienced by the patient. To do this, we will test the hypotheses that a) those patients with greater mobilization and visitation rates and decreased anxiety and pain levels will have a greater self-perceived readiness for discharge and b) that patients who receive daily mobilization goals and personal motivation will have higher step rates, and therefore have a greater self-perceived readiness for discharge, than those that do not.

Ninety-nine patients will be recruited to participate in this intervention-based study. Patients will be identified by the surgeons as potential participants, and referred to the study coordinator. The study coordinator will obtain informed signed consent after the patient's physician appointment in the clinical offices. At this point, participant medical information will be collected and participants will be asked to complete the EORTC QLQ C-30 Quality of Life (QOL) questionnaire. Participants will then be randomly assigned to one of three intervention groups. The intervention groups are: G0 (no intervention), G1 (minimal intervention) and G2 (maximal intervention). Participants in the G0 group will receive the standard clinical care outlined in the present nursing clinical pathway sheets, including a pre-operative video on what to expect post-operatively. G1 participants will receive the same standard clinical care as G0 patients, but will also receive a personal ambulation goal sheet and log book to help them monitor their rate of mobility and their achievement of daily goals. G2 participants will receive the same care as G1 patients, but will also receive a daily visit from the study coordinator to help them monitor their physical activity and motivate them to achieve their goals.

Patients from all levels of intervention will fill out a questionnaire (T.R.I.M Readiness for Discharge Questionnaire, titled T.R.I.M. Participant Questionnaire when handed to participants) on their pain, anxiety and their self-perceived readiness for discharge on post-operative days 3 and 5, day of discharge and on their follow-up visit. The T.R.I.M Readiness for Discharge Questionnaire contains the Short Form - McGill Pain Questionnaire [Melzack, 1987], the Short Form State-Trait Anxiety Index [Marteau & Bekker, 1992]. Moreover, the questionnaire asks the patient about their self-perceived readiness for discharge. They are asked to answer the question "Are you ready to go home?" by marking an X on a line (a visual analog scale, VAS) where one end of the line indicates "Not at all" and the other "Definitely". Patients will also be instructed to have their visitors sign-in and -out on a log sheet and be outfitted with a pedometer to measure the number of steps they take in a day. Also on the day of discharge, patients will be asked to fill out the EORTC Quality of Life questionnaire again. Finally, 1 month after discharge patients will be contacted for follow up and to complete the EORTC questionnaire a third time along with the Participant Questionnaire. All individuals will be visited daily by the study coordinator while they are in the hospital, who will record their daily steps. During these daily visits, the study coordinator will also examine the goals of the participants in the G2 intervention group. They will be verbally encouraged to meet their ambulation goals. Those in the G0 and G1 intervention groups will only have their daily steps recorded.

T-tests and Chi-Square analysis will be used on means and proportions respectively, to determine any differences between the intervention groups. Logistic regression analysis will be carried out and Pearson's correlation coefficients will be calculated to examine the factors that contribute to a patient's self-perceived readiness for discharge, their post-operative Quality of Life and their length of stay. Multivariate analysis of variance will be used on ambulation rates, visitation rates, pain scores, anxiety scores and readiness for discharge to examine differences between the different interventions and other factors describing the patient's clinical pathway (i.e. length of stay, days on analgesics, and hospital costs/patient).

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective lobectomy,
* speak, write and read English,
* ambulate prior to surgery

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2005-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Perceived readiness for discharge VAS score (at discharge)

SECONDARY OUTCOMES:
Length of stay, physician's and nurses perceived readiness for discharge, visitation rates, anxiety score, pain score (at discharge), primary and secondary outcomes (at post-op days 3, 5 and follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: John Yee, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital Chest Centre, Vancouver, British Columbia, Canada